CLINICAL TRIAL: NCT04063800
Title: Prediction of the Risk of Biochemical Relapse After Radical Prostatectomy for Prostate Cancer Using Radomics on Pre-therapeutic MRI
Acronym: PREBOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PREBOP (29BRC18.0108)
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Prostatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With 50% of post-operative biochemical failure, efficient predictive models are needed to guide post-operative management.

Radiomic features are quantitative features extracted from medical imaging, supposed to be correlated with tumor heterogeneity.

We aim to build and test three predictive models (clinical, radiomic and combined models).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18yo
* Patients underwent radical prostatectomy
* High-risk prostate cancers: at least 1 criteria (pt3a/pT3b/pT4, R1, Gleason score > 7)

Exclusion Criteria:

* No available pre-operative MRI
* No analyzable pre-operative MRI
* proof of lymph-node involvement (cN1/2 or pN1/2)
* post-operative PSA > 0.04ng/mL

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Study Population: - Patients with high-risk prostate cancers who underwent pre-operative prostate MRI followed by radical prostatectomy +/- lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Prediction of biochemical failure | From the date of surgery until data collection (up to 100 months)
  Comparison of AUCs between each predictive model

SECONDARY OUTCOMES:
Prediction of survival without biochemical failure | From the date of surgery until data collection (up to 100 months)
  Survival analysis: comparison of Kaplan-Meier curves

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest, Brittany Region
  - Centre Hospitalier de Cornouaille, Quimper, Brittany Region

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.